CLINICAL TRIAL: NCT02368587
Title: Randomised, Double-blind, Placebo-controlled, Intracoronary or Intravenous Infusion Human Wharton' Jelly-derived Mesenchymal Stem Cells in Patients With Ischemic Cardiomyopathy
Brief Title: Intracoronary or Intravenous Infusion Human Wharton' Jelly-derived Mesenchymal Stem Cells in Patients With Ischemic Cardiomyopathy
Acronym: WJ-ICMP Tria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: First People's Hospital of Foshan (Other); General Hospital of Armed Police, Beijing (Unknown); PLA General Hospital, Beijing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NavyGHB
Record Dates: First submitted 2015-02-03; First posted 2015-02-23 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Cardiomyopathy
Keywords: intracoronary infusion; intravenous infusion; Wharton's jelly-derived mesenchymal stem cells; ischemic Cardiomyopathy; heart function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracoronary infusion WJMSCs (Placebo Comparator): Intracoronary infusion WJMSCs or placebo in patients with ischemic heart failure
  Interventions: Biological: WJMSCs Vs. placebo
- Intravenous infusion WJMSCs (Placebo Comparator): Intravenous infusion WJMSCs or placebo in patients with ischemic heart failure.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: WJMSCs Vs. placebo — WJMSCs Vs. placebo
  Arms: Intracoronary infusion WJMSCs
Biological: Placebo — WJMSCs Vs. placebo
  Arms: Intravenous infusion WJMSCs

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of intracoronary or intravenous infusion human umbilical Wharton's jelly-derived Mesenchymal Stem Cell (WJMSC) in patients with ischemic cardiomyopathy secondary to myocardial infarction.

DETAILED DESCRIPTION:
Ischemic heart failure (IHF) secondary to myocardial infarction is a common, lethal, disabling, and expensive condition. Despite advances over the last 30 years, the prognosis of patients with IHF remains poor. At present, there has been increasing interest in attempting to repair the failing heart with the use of stem cells, since this approach has the potential to regenerate dead myocardium and thus alleviate the underlying cause of IHF.

A very primitive population of mesenchymal stem cells (MSCs) has been isolated from a continuum from the sub-amnion to perivascular region of umbilical cord, referred to as Wharton's jelly-derived MSCs (WJMSCs). WJMSCs retain a combination of most of their embryonic stem cell (ESC) and MSC markers in primary culture and early passages, thus retaining their multipotent stem cell characteristics. Preclinical studies have demonstrated that WJMSCs can be induced to differentiate into cardiomyocytes and endothelial cells and to integrate into the vasculature and ischemic cardiac tissue, as well as to improve heart function significantly. Therefore, the investigators performed a double-blind, placebo-controlled trial, randomly assigning 160 patients with ischemic heart failure secondary to myocardial infarction to receive an intracoronary or intravenous infusion of WJMSCs or placebo, to investigate the therapeutic safety and efficacy of WJMSCs in patients with ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age no limited
2. Patient must provide written informed consent.
3. Have a diagnosis of chronic ischemic left ventricular dysfunction secondary to myocardial infarction (MI) as defined by any of the following 3 criteria:

   * Previous MI is documented by a clinical history that includes an elevation of cardiac enzymes and/or electrocardiogram (ECG) changes consistent with MI.
   * Patients treated with thrombolytic therapy or percutaneous coronary revascularization.
   * Screening CMRI shows an area of akinesis, dyskinesis, or severe hypokinesis associated with evidence of myocardial scarring based on delayed hyperenhancement after gadolinium infusion.
4. Patient has been treated with appropriate maximal medic al therapy for ICMP. For β -blockade, the patient must have be en on a stable dose of a clinically appropriate β-blocker for 3 months. For angiotensin-converting enzyme inhibition, the patient must have been on a stable dose of a clinically appropriate agent for 1 m
5. left ventricular ejection fraction (LVEF)<45% by echocardiogram, CMRI, or left ventriculogram within the prior 6 m
6. Patients who are a candidate for cardiac catheterization assignment intracoronary infusion group; but patients in no-candidate for cardiac catheterization assignment intravenous infusion group.

Exclusion Criteria:

1. Have a baseline glomerular filtration rate > 50 mL/min per 1.73 m2
2. Evidence of a life-threatening arrhythmia (ventricular tachycardia or complete heart block) on screening ECG..
3. Have a hematologic abnormality as evidenced by hematocrit <25% , white blood cell <2500/u L or platelet values<100000/u L without another explanation.
4. Have liver dysfunction , as evidenced by enzymes (aspartate aminotransferase and alanine aminotransferase) >3× the upper limits of normal.
5. Have a coagulopathy (international normalized ratio > 1.3) not because of a reversible cause (ie, coumadin).
6. Have a contraindication to performance of CMRI (CMRIs will be performed in patients with pacemaker who are not pacemaker dependent).
7. Be an organ transplant recipient.
8. Have a clinical history of malignancy within 5 y except curatively treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
9. Have a noncardiac condition that limits lifespan to <1y.
10. Have a history of drug or alcohol abuse within the past 24 m.
11. Be serum positive for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C.
12. Be a female who is pregnant, nursing, or of childbearing potential who is not practicing effective contraceptive methods.

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The primary end point was safety in incidence of adverse events (AEs) within 12 months | 12 months
  the incidence of adverse events (AEs) within 12 months, including death, nonfatal MI, stroke, hospitalization for worsening heart function, severe arrhythmias, repeated coronary intervention, stent thrombosis, coronary artery microvascular obstruction, immune system disorders, or ectopic tissue formation, was monitored and quantified. Laboratory assays, including biochemical assays, hematologic, tumor and immune indexes and Holter monitoring, were performed at the different follow-up times at 1 months-1 year. The trial will be monitored by a Data and Safety Monitoring Board (DSMB) and the trial will be discontinued in case of safety concerns.

SECONDARY OUTCOMES:
The secondary end point was efficacy in absolute change of the global LV ejection fraction (LVEF) from baseline to 12 months by MRI | 12 months
  The secondary end point was efficacy, which was assessed in terms of the absolute change in the global LV ejection fraction (LVEF) from baseline to 12 months post-treatment, as measured by cardiac magnetic resonance imaging (CMRI). Furthermore, CMRI assessments measured scar mass and viable myocardial mass in the left ventricle, scar size, cardiac volumes, global function, regional function, and 6-min walk tests in all patients from baseline to 12 months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ning K Zhang, MS, Study Director — Navy General Hospital, Beijing